CLINICAL TRIAL: NCT06391996
Title: Genetics-based Efficacy Analysis: Ustekinumab Versus Secukinumab for the Treatment of Generalized Pustular Psoriasis
Brief Title: Biologic Therapy for Generalized Pustular Psoriasis
Status: Completed | Type: Observational
Sponsor: Chao Ji (Other)
Responsible Party: Sponsor-Investigator, Chao Ji, Head of dermatology, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: MRCTA,ECFAH of FMU [2022]007
Record Dates: First submitted 2024-04-20; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Generalized Pustular Psoriasis
Keywords: Secukinumab; Ustekinumab; Clinical efficacy; Generalized pustular psoriasis; Safety; Gene mutations
MeSH Terms: conditions — Psoriasis | interventions — Genotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- the ustekinumab group: Before treatment, participants underwent routine blood and urine tests, erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), liver and kidney function tests, tuberculous infection of T cells spot tests, hepatitis B virus marker tests, chest CT scans, etc. After exclusion of relevant contraindications, participants received subcutaneous ustekinumab therapy. During the treatment period, participants received ustekinumab at weeks 0, 4, 16, and every 12 weeks thereafter until week 48. The single dose of ustekinumab was 45 mg for adult subjects weighing ≤ 100 kg, and 90 mg for subjects weighing > 100 kg. The ustekinumab dosage for pediatric participants was 0.75 mg/kg for participants weighing < 60 kg; 45 mg for pediatric participants weighing 60 kg to 100 kg; and 90 mg for pediatric participants weighing > 100 kg.
  Interventions: Drug: After exclusion of relevant contraindications, participants received subcutaneous ustekinumab/secukinumab therapy.
- the secukinumab group: Before treatment, participants underwent routine blood and urine tests, erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), liver and kidney function tests, tuberculous infection of T cells spot tests, hepatitis B virus marker tests, chest CT scans, etc. After exclusion of relevant contraindications, participants received subcutaneous secukinumab therapy. During the treatment period, participants received secukinumab at weeks 0, 1, 2, 3, and 4, and every 4 weeks thereafter until week 48. The secukinumab dosage was 300mg for adult humans. Pediatric participants received a dose based on their weight category (< 50 kg, ≥ 50 kg): participants weighing < 50 kg received 75 mg, those weighing ≥ 50 kg received 150 mg.
  Interventions: Drug: After exclusion of relevant contraindications, participants received subcutaneous ustekinumab/secukinumab therapy.

INTERVENTIONS:
Drug: After exclusion of relevant contraindications, participants received subcutaneous ustekinumab/secukinumab therapy. — During the treatment period, participants received either ustekinumab at weeks 0, 4, 16, and every 12 weeks thereafter until week 48, or secukinumab at weeks 0, 1, 2, 3, and 4, and every 4 weeks thereafter until week 48. The dose of ustekinumab/secukinumab was referenced to the dose used for moderate to severe plaque psoriasis. The single dose of ustekinumab was 45 mg for adult subjects weighing ≤ 100 kg, and 90 mg for subjects weighing > 100 kg. The ustekinumab dosage for pediatric participants was 0.75 mg/kg for participants weighing < 60 kg; 45 mg for pediatric participants weighing 60 kg to 100 kg; and 90 mg for pediatric participants weighing > 100 kg. The secukinumab dosage was 300mg for adult humans. Pediatric participants received a dose based on their weight category ( <50 kg, ≥50 kg): participants weighing < 50 kg received 75 mg, those weighing ≥ 50 kg received 150 mg.
  Other Names: The investigators collected participants' saliva for genotyping.

SUMMARY:
The investigators aim to compare the efficacy and safety of secukinumab and ustekinumab in patients with generalized pustular psoriasis (GPP), and to explore the impact of genetic mutation types on clinical efficacy. The main questions the study aims to answer are:

Is there a difference in the effectiveness of secukinumab and ustekinumab in the treatment of GPP? How is the safety of secukinumab and ustekinumab in the treatment of GPP? Does the type of genetic mutation in GPP patients affect the efficacy of secukinumab and ustekinumab? The investigators will compare patients treated with secukinumab to those treated with ustekinumab to see the difference in the effectiveness of the two drugs in treating GPP.

Participants will:

The investigators conducted a 48-week follow-up study on 65 participants who were admitted to the dermatology department of the First Affiliated Hospital of Fujian Medical University for GPP from July 2019 to December 2022. All participants underwent saliva-based genetic testing.

Efficacy analyses were performed based on the scores of Generalized Pustular Psoriasis Area and Severity Index (GPPASI) and Generalized Pustular Psoriasis Physician Global Assessment (GPPGA) at week 0, 2, 4, 12, 24, and 48.

Participants were also asked to report all adverse events (AEs) during follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meet the diagnostic criteria for GPP.
2. Patients had an average GPPGA score of 3 or higher (moderate to severe disease).
3. Patients had discontinued the treatment with non-biologic agents before they started the treatment with ustekinumab/secukinumab.

Exclusion Criteria:

1. Pregnant and lactating patients.
2. Patients with malignant tumors.
3. Patients with a history of multiple drug allergies or a severe allergic constitution.
4. Contraindications for ustekinumab/secukinumab, including active tuberculosis, active hepatitis B, hepatitis C, or inflammatory bowel disease.

Patients who were severely immunocompromised.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a retrospective study of adult and pediatric patients with GPP. The investigators obtained data for 65 patients (33 children, 32 adults) who were admitted to the Department of Dermatology in the First Affiliated Hospital of Fujian Medical University because of GPP between July 2019 and Dec 2022. All patients were followed for 48 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
To compare the clinical efficacy difference between ustekinumab and secukinumab in the treatment of GPP through evaluation of GPPASI. | 48 weeks
  Efficacy analyses were performed based on the scores of Generalized Pustular Psoriasis Area and Severity Index (GPPASI) at week 0, 2, 4, 12, 24, and 48. GPPASI provided a numeric scoring system to assess patient's overall disease state of GPP, ranging from 0 to 72, with higher scores indicating more severe conditions. Clinical efficacy was evaluated by GPPASI -50, -75, -90, and -100 responses at each time point.

SECONDARY OUTCOMES:
To compare the clinical efficacy difference between ustekinumab and secukinumab in the treatment of GPP through evaluation of GPPGA. | 48 weeks
  Efficacy analyses were performed based on the scores of Generalized Pustular Psoriasis Physician Global Assessment (GPPGA) at week 0, 2, 4, 12, 24, and 48. The investigator scored the erythema, pustules, and scale of all GPP lesions from 0 to 4 using GPPGA. Each component was graded separately, and the average was calculated. The final GPPGA was determined by this composite score.
By saliva-based genetic testing, analyze the mutation rates of common mutation gene sites in GPP. | 48 weeks
  To analyze whether gene mutations cause different responses to ustekinumab and secukinumab in GPP patients.
Analyzing the incidence of adverse reactions to ustekinumab and secukinumab in the treatment of GPP. | 48 weeks
  During the follow-up period, participants are requested to report all adverse reactions experienced since their last visit, such as rash, diarrhea, infections, etc., and record the type, onset time, severity, duration, triggering, and relieving factors of the adverse reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China